CLINICAL TRIAL: NCT05099081
Title: Effectiveness of Diode Laser Versus Sclerotherapy in the Treatment of Oral Pyogenic Granuloma: a Randomized-controlled Clinical Trial
Brief Title: Effectiveness of Diode Laser and Sclerotherapy in Treatment of Oral Pyogenic Granuloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0008839
Record Dates: First submitted 2021-09-09; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Pyogenic Granuloma of Gingiva
Keywords: Pyogenic granuloma; Diode laser; Sclerotherapy; Ethanolamine oleate
MeSH Terms: conditions — Granuloma, Pyogenic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- diode laser (Experimental): diode laser application
  Interventions: Procedure: diode laser application
- sclerotherapy (Active Comparator): intra-lesional injection of ethanolamine oleate
  Interventions: Procedure: intra-lesional injection of ethanolamine oleate

INTERVENTIONS:
Procedure: diode laser application — Local anesthesia will be applied Lesion will be excised with diode laser (Medency, Italy) continuous wave mode 980 nm wave length with an output power 3 W in contact mode
  Arms: diode laser
Procedure: intra-lesional injection of ethanolamine oleate — Local anesthesia will be applied Injection of ethanolamine oleate (sclerosing gent) with concentration 5% diluted in distilled water to form 2.5% ethanolamine oleate According to lesion size range from 1.5 to 3 ml of solution will be injected slowly into lesion using gauge needle until leaked from lesion.
  Lesion will be compressed for 5 minutes. Lesion will be observed once a week after injection until it becomes necrotic and falls off spontaneously.
  Repeated injection may be needed.
  Arms: sclerotherapy

SUMMARY:
To clinically assess the effectiveness of diode laser versus sclerotherapy in the treatment of oral pyogenic granuloma.

A randomized-controlled clinical trial conducted on 20 patients with oral pyogenic granuloma. Patients were assigned into two groups. Group I treated by diode laser1; group II treated by injection of ethanolamine oleate2 as sclerosing agent. All patients were clinically assessed for pain, bleeding during surgery and healing quality; 1st week, 2nd week and 4th week. The patients were followed up after 3 months from the end of treatment.

DETAILED DESCRIPTION:
Background: Pyogenic granuloma (PG) is one of the most common reactive hyperplasia that causes soft tissue enlargement. It affects skin and oral mucosa. The traditional treatment for oral PG is conservative surgical excision with cold blade together with the removal of causative irritant or source of trauma. Bleeding susceptibility, healing quality and pain represent common complications following surgical excision of pyogenic granuloma. Sclerosing agents are widely used in the treatment of pyogenic granuloma as it is a conservative non painful procedure. The use of lasers in dentistry have grown in the last 4 decades. It has proved its efficacy in the treatment of pyogenic granuloma.

Study objective: Study will be conducted to evaluate healing quality of using diode laser versus sclerotherapy (Ethanolamine oleate) in the treatment of oral pyogenic granuloma.

Materials and Method: This randomized controlled clinical trial will include 20 patients with pyogenic granuloma, divided equally into two groups. Group-I (test group) will be managed by application of diode laser. Group- II (control group) will be managed by injection of ethanolamine oleate as sclerosing agent on weekly injection visits. Patients of both groups will be evaluated intraoperatively for bleeding severity and postoperatively in terms of pain at the 2nd and 7th day and healing quality.

Results: Results will be tabulated and statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders diagnosed clinically and confirmed histologically with oral pyogenic granuloma.
2. Size of the lesion not less than 5mm.
3. Patients included in the study will be having gingival pyogenic granuloma as it is the most common site for its occurrence.
4. Patient age ranges from 19 to 50 years old.

Exclusion Criteria:

1. Patients with uncontrolled diabetes.
2. Immuno-compromised patients.
3. Patients with renal disease.
4. Patients having coagulation disorders.
5. Patients having allergic reaction to any of the sclerosing drug constituents.
6. Pregnant and lactating women.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Bleeding | at baseline
  Mild: Subsides at 20 min after applying pressure with gauze. Moderate: Requires haemostatic irrigation. Severe: Needs suturing and might need vitamin K administration or fresh frozen plasma infusion.
Change in pain score | at 2nd and 7th day
  Postoperative pain will be evaluated at 2nd and 7th day using numeric rating scale (NRS) 0 = no pain. 1-3 = mild pain. 4-6 = moderate pain. 7-10 = severe pain.
Change in healing quality index | at 1st week, 2nd week ,4th week and 3rd month
  Will be measured according to landry classification
  1. = very poor
  2. = poor
  3. = good
  4. = very good
  5. = excellent

CONTACTS AND LOCATIONS:
Overall Officials: Sandra N. Edward, B.D, Principal Investigator — Alexandria University
Locations (1):
- Faculty of dentistry, Alexandria University, Alexandria, Egypt